CLINICAL TRIAL: NCT01977638
Title: Phase 1 Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CXD101 Given Orally (Twice Daily Dosing for 5 Consecutive Days in a 21-day Period) in Patients With Advanced Malignancies Expressing the Biomarker HR23B
Brief Title: Phase 1 Trial of CXD101 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other); National Institute for Health Research, United Kingdom (Other Government); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXD101-0901; 2009-012743-42 (EudraCT Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-07 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2021-10

CONDITIONS: Advanced Cancer
Keywords: Advanced solid tumours; Lymphoma; Myeloma
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CXD101 (Experimental): Dose escalation study of CXD101 administered orally twice daily for 5 consecutive days in every 21 day cycle. Starting dose 1mg twice daily (2mg/day).
  Interventions: Drug: CXD101

INTERVENTIONS:
Drug: CXD101 — Capsules, administered orally
  Other Names: AZD9468

SUMMARY:
The purpose of this study is to determine the highest dose of CXD101 (a novel histone deacetylase inhibitor) that can be safely administered to patients with advanced tumours. The study will also investigate the use of HR23B expression in tumour as a biomarker of response to treatment with CXD101. Patients with solid tumours, lymphoma and myeloma can be considered for this study.

DETAILED DESCRIPTION:
Patients will be treated with CXD101 administered orally starting at 1mg twice a day (ie: 2mg/day). Dose escalation will proceed according to a standard 3+3 phase 1 scheme. Adverse experiences will be evaluated according to the NCI Common Terminology Criteria for Adverse Events, version 4.0. Dose escalation will continue until dose limiting toxicity is encountered in >1/3rd of patients at any dose level. The dose level below this will be determined to be the maximum tolerated dose. Patients will be treated, at the discretion of the Principal Investigator, until disease progression, unacceptable toxicity or the withdrawal of consent. At the maximum tolerated dose a further 20 patients, defined by tumour HR23B expression will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Life expectancy of at least 12 weeks.
3. ECOG performance score of ≤ 1
4. Histologically or cytologically confirmed malignant tumour with the potential to benefit from HDAC inhibitor therapy.
5. High HR23B expressing tumour sample on IHC (expansion cohort only).
6. Evaluable disease.
7. The patient is willing and able to comply with the protocol for the duration of the study, including scheduled follow-up visits and examinations.
8. Patients must have recovered from effects of prior treatments, including surgeries (persistent grade 1 toxicities are permitted at the discretion of the Chief Investigator).
9. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 14 days prior to start of trial. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 16 weeks after discontinuation of treatment. Oral contraception and parenteral hormonal contraceptives (patches, injectables and implants) that may be affected by enzyme-inducing drugs should only be used in combination with a barrier method. All males with partners of childbearing potential or whose partners are pregnant must use barrier contraception for the duration of dosing and for 16 weeks post-dosing.
10. Able to give written (signed and dated) informed consent.
11. Haematological and biochemical indices within acceptable ranges as detailed in study protocol.

Exclusion Criteria:

1. Pregnant or breast-feeding women or women of childbearing potential unless effective methods of contraception are used.
2. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
3. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.
4. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or use of other investigational agents within 28 days prior to trial entry (or a longer period depending on the defined characteristics of the agents used). Limited field radiotherapy to an isolated lesion in bone or soft tissue must be completed 2 weeks prior to trial entry.
5. Patients must not receive any concurrent anti-cancer therapy, including investigational agents, while on-study. Patients may continue the use of bisphosphonates for bone disease or corticosteroids providing the dose is stable before and during the trial.
6. Major surgery within 4 weeks of starting the study.
7. Co-existing active infection requiring parenteral antibiotics or serious concurrent illness deemed clinically significant.
8. Patients with known brain metastases, unless these are shown to be stable (symptomatically and/or radiologically) over a period of 2 months or more.
9. History of refractory nausea and vomiting, chronic GI diseases (eg: inflammatory bowel disease) or significant bowel resection that would preclude adequate absorption of oral medication.
10. Patients who are unable to swallow oral medication.
11. Patients with corrected QT interval >450msec.
12. Persistent grade 2 or greater toxicities from any cause.
13. Previous treatment with a HDAC inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of CXD101 administered twice daily for 5 consecutive days every 21 days | 18 months

SECONDARY OUTCOMES:
To determine the pharmacokinetic (PK) profile of CXD101 following single and multiple dosing | 18 months
To enable a preliminary assessment of the anti-tumour activity of CXD101 | 24 months
To evaluate the tissue expression of the biomarker HR23B | 24 months
To assess the pharmacodynamic effect of CXD101 | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth SW, Eyre TA, Whittaker J, Campo L, Wang LM, Soilleux E, Royston D, Rees G, Kesavan M, Hildyard C, Kazmi F, La Thangue N, Kerr D, Middleton MR, Collins GP. A Phase 2a cohort expansion study to assess the safety, tolerability, and preliminary efficacy of CXD101 in patients with advanced solid-organ cancer expressing HR23B or lymphoma. BMC Cancer. 2021 Jul 23;21(1):851. doi: 10.1186/s12885-021-08595-w. PMID 34301221